CLINICAL TRIAL: NCT03234894
Title: Clinical Study of the WoundCare360 SiteSeal Adjunctive Compression Device Following Interventional Endovascular Procedures
Brief Title: Clinical Trial of the WC360 SiteSeal Adjunctive Compression Device Following Interventional Endovascular Procedures
Acronym: SiteSeal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wound Care 360, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G150106/A001
Record Dates: First submitted 2016-06-28; First posted 2017-07-31 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SiteSeal Endovascular (Other): After intervention (deployment and removal of the Site Seal endovascular adjunctive compression device), the physician determines whether or not there was laceration of the femoral nerve or laceration of the femoral artery per protocol. A series of possible minor and/or major complications are noted per protocol.
  There is a secondary metric as to patient reported pain on a 1-10scale.
  Interventions: Device: SiteSeal Endovascular

INTERVENTIONS:
Device: SiteSeal Endovascular — to evaluate the safety of the SiteSeal™ Endovascular Adjunctive Compression Device across a broad array of patients undergoing interventional endovascular procedures.
  Other Names: SiteSeal Cardiovascular

SUMMARY:
This Clinical Study is a pivotal study to evaluate the safety of the SiteSeal™ Adjunctive Compression Device across a broad array of patients undergoing interventional endovascular procedures.

DETAILED DESCRIPTION:
The study design is a single arm with 90 patients. The primary endpoints measure the risk for common femoral nerve damage and common femoral artery laceration from the blind placement of a Z-stitch in the soft tissue above the femoral bundle.

The sample size is 90 patients. The project objective is to demonstrate the safety of the device.

ELIGIBILITY:
Inclusion Criteria

1. Patients between the ages 19 to 90
2. Patient or his/her legally authorized representative, has given written informed consent for participation prior to the procedure
3. Procedure is an interventional procedure
4. Patient is willing to undergo all study procedures and adhere to data collection and follow-up requirements
5. Patient is a candidate for elective, non-emergent cardiac or peripheral vascular catheterization from the femoral artery approach
6. Patient is willing to have a pre/post procedure ultrasound.

Exclusion Criteria:

1. Patients are <19 years old
2. Patients are >90years old
3. Patient has received GP IIb/IIIa inhibitors
4. Patient or patient's representative is unable to provide written informed consent.
5. Patient is unable or unwilling to adhere to data collection and follow-up requirements
6. Procedure is emergency PCI
7. Patient is on dialysis
8. Patient has a known diagnosis of fibromyalgia
9. Patients with acute coronary syndrome (i.e., unstable angina or myocardial infarction) ≤ 48 hours before this catheterization procedure.
10. Patients with systolic blood pressure < 90 mm Hg at the end of the catheterization procedure
11. Patients who are immunocompromised
12. Patients with preexisting systemic infection or local infections at the access site
13. Patients who are known or suspected to be pregnant, or are lactating
14. Patients who have undergone prior or recent use of an intra-aortic balloon pump through the arterial access site above the inguinal ligament
15. Patients who have undergone prior vascular closure device use in the ipsilateral common femoral artery ≤ 30days before this catheterization procedure
16. Patients who have undergone prior use of manual or mechanical compression for closure in the ipsilateral common femoral artery ≤30 days before the catheterization procedure
17. Patients requiring a repuncture at a site previously punctured within 48 hours of the catheterization procedure
18. Patients who have undergone an antegrade puncture
19. Patients with puncture sites believed to be in the profunda femoris artery, superficial femoral artery, or at the bifurcation of these arteries
20. Patients with puncture tract angle >55°
21. Patients who are suspected to have experienced a femoral artery back wall puncture or who underwent > 1femoral artery puncture during the catheterization procedure
22. Patient with significant anemia (hemoglobin < 10 g/dL, Hct < 30%)
23. Patients with a known bleeding disorder, including thrombocytopenia (platelet count < 100,000 cells/μL), thrombasthenia, hemophilia, or von Willebrand's disease
24. Patients with systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg at the end of this catheterization procedure, unless systolic and/or diastolic pressure was lowered by pharmacological agents prior to the end of the catheterization procedure
25. Patients with a baseline INR >1.5 (e.g., on warfarin therapy)
26. Patients whose ACT >300seconds at the end of the catheterization procedure
27. Patients who have undergone administration of low molecular weight heparin (LMWH) within 8hours of this catheterization procedure
28. Patients in whom continued heparin or other anticoagulant/antiplatelet therapy is planned for this patient (with the exception of glycoprotein IIb/IIIa inhibitor therapy) during the first few hours following the catheterization procedure
29. Patients having a complication or complications at the femoral artery access site during the catheterization procedure including bleeding, hematoma, intraluminal thrombus, pseudoaneurysm, or arteriovenous fistula
30. Patients with an ipsilateral or bilateral lower extremity amputation(s)
31. Patient known to require extended hospitalization (e.g., patient is undergoing cardiac surgery)
32. Patients who have a planned endovascular procedure within the next 30days after the catheterization procedure
33. Patients who are currently participating in another investigational study that has not concluded the follow-up period
34. Patients who have already participated in the IDE study
35. Patients who cannot adhere to or complete the study for any reason including but not limited to geographical residence or life-threatening disease

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
The percent of patients with common femoral nerve damage or with bleeding from femoral artery laceration from the blind placement of a Z-stitch in the soft tissue above the femoral bundle. | 24 hours
  Femoral damage is indicated if the patient has an audible response during suture placement. Arterial laceration is visible bleeding during suture placement.

SECONDARY OUTCOMES:
Patient-rated patient discomfort. | 24 hour interview
  Patients are called back after 24 hours and asked to rate their discomfort on a 1-10 scale. The mean of all patients 1-10scale rating is reported as the discomfort of the arm.
The percent of patients who had a major complication. | 30day interview
  Major complications are defined in the protocol. Major complications are summed and the mean of the entire arm is reported as a percent of patients who had major complications.
The percent of patients who had a minor complication. | 30day interview
  Minor complications are defined in the protocol. Minor complications are summed and the mean of the entire arm is reported as the percent of patients who had minor complications.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Kassab, MD, Principal Investigator — MOVI; Matthew Earnest, MD, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT03234894/SAP_000.pdf
  • Study Protocol (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03234894/Prot_001.pdf
  • Informed Consent Form (2015-04-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03234894/ICF_002.pdf